CLINICAL TRIAL: NCT05719714
Title: Effect of Dapagliflozin on Metabolomics and Cardiac Mechanics in Chronic Kidney Disease
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Rupal Mehta, Doctor of Medicine, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STU00215566; K23HL150236 (NIH)
Record Dates: First submitted 2023-01-31; First posted 2023-02-09 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Chronic Kidney Diseases; Heart Failure With Preserved Ejection Fraction; Kidney Diseases; Heart Failure
Keywords: kidney; heart failure; kidney diseases
MeSH Terms: conditions — Renal Insufficiency, Chronic; Kidney Diseases; Heart Failure | interventions — dapagliflozin

STUDY DESIGN:
Intervention Model Description: 30 subjects will be randomized to intervention. 30 subjects will be randomized to standard of care.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Intervention group (Experimental): Thirty individuals will be randomized to dapagliflozin 10mg to be taken daily for six months.
  Interventions: Drug: Dapagliflozin 10 MG [Farxiga]
- Standard of Care group (No Intervention): Thirty individuals will be randomized to standard of care treatment.

INTERVENTIONS:
Drug: Dapagliflozin 10 MG [Farxiga] — 10mg (milligram) tablet to be taken orally once daily for 6 months. Manufacturer: Astrazeneca. Study drug will be stored and dispensed by the Interventional Drug Service Pharmacy at Northwestern University.
  Arms: Intervention group

SUMMARY:
The goal of this study is to better understand the effects of a sodium-glucose transport protein 2 inhibitor, dapagliflozin, added on to standard of care on heart and lung function and circulating metabolites (substances created when our bodies break down food, drugs, or its own tissues) in patients with chronic kidney disease.

DETAILED DESCRIPTION:
This is a 6-month interventional patient-oriented research study of sixty patients with chronic kidney disease (CKD) and evidence of subclinical heart failure with preserved ejection fraction (HFpEF) (estimated glomerular filtration rate [eGFR] 25-60 ml/min/1.73m2, absolute left ventricular longitudinal strain [LVGLS] <18% or left atrial reservoir strain (LARS) < 25% on 2D-speckle tracking echocardiography or meeting 3/5 of the American Society of Echocardiography criteria for diastolic dysfunction: septal e' <7 cm/sec, lateral e'<10 cm/sec, average E/e' ratio>14, left atrial volume index >34 mL/m2, or peak tricuspid regurgitation velocity >2.8 m/sec), or peak VO2 Females: ≤ 18 mL/kg/min, peak VO2 Males: ≤ 20 mL/kg/min on cardiopulmonary exercise testing, or lack of augmentation of LVLS or LARS during exercise. Half of the patients will be randomized to receive dapagliflozin for six months as an add-on to standard of care (SOC). Metabolomic testing and cardiac and functional exercise testing will be done at baseline and at six months. The aim of the current study is to investigate whether SGLT2i-induced metabolomic changes are associated with improved cardiac and functional testing ascertained on 2D-speckle tracking echocardiography or cardiopulmonary functional testing at six months.

ELIGIBILITY:
Inclusion Criteria:

1. >18 years of age
2. eGFR 25-60 ml/min/1,73m2 (eGFR = estimated glomerular filtration rate)
3. On stable doses of diuretics and/or angiotensin converting enzyme inhibitor or angiotensin receptor blocker
4. Evidence of subclinical heart failure with preserved ejection fraction at their pre-exercise echocardiogram (defined as meeting 3/5 of the American Society of Echocardiography (ASE) criteria for diastolic dysfunction [septal e'<7 cm/wc, average E/e' ratio>14, left atrial volume index >34 mL/m2, and peak TR velocity >2.8 m/sec] or absolute left ventricular longitudinal strain < 18%, left atrial reservoir strain (LARS) < 25% on 2d speckle tracking echocardiography), lack of augmentation of LVLS or LARS during exercise, or peak VO2 Females: ≤ 18 mL/kg/min, peak VO2 Males: ≤ 20 mL/kg/min on cardiopulmonary exercise testing.

Exclusion Criteria:

1. presence or history of diabetes
2. coronary revascularization within the last 6 months
3. hemodynamically significant valvular disease
4. significant lung disease requiring home oxygen
5. angina (chest pain)
6. non-revascularized myocardial ischemia
7. systolic BP <100 or >180 mmHg
8. pregnancy
9. clinical heart failure symptoms
10. history of systemic disease processes that can cause HFpEF such as amyloidosis or sarcoidosis
11. any musculoskeletal or chronic condition that will interfere with completion of cardiac testing
12. active cancer
13. immunosuppressive therapy
14. baseline or pre-exercise echocardiogram demonstrates a reduced ejection fraction < 50%
15. currently on sodium glucose cotransporter 2 inhibitor (SGLT2i) therapy
16. Hypersensitivity to a SGLT2i
17. Pre-existing liver disease
18. ALT/AST> 3x normal (ALT = alanine aminotransferase AST = aspartate aminotransferase)
19. history of recurrent urinary tract infections (in the opinion of the investigator) or a urinary tract infection in the last 3 months

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-01-16 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Left ventricular longitudinal strain (LVLS) | 6 months
  2D-speckle tracking echocardiography
Peak VO2 (oxygen consumption) | 6 months
  Cardiopulmonary exercise stress test
Circulating plasma metabolite concentrations | 6 months
  Plasma

SECONDARY OUTCOMES:
Left Atrial Reservoir Strain (LARS) | 6 months
  2D-STE
Right ventricular free wall strain | 6 Months
  2D-STE

CONTACTS AND LOCATIONS:
Overall Officials: Rupal Mehta, MD, Principal Investigator — Northwestern Univeristy
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Benjamin EJ, Virani SS, Callaway CW, Chamberlain AM, Chang AR, Cheng S, Chiuve SE, Cushman M, Delling FN, Deo R, de Ferranti SD, Ferguson JF, Fornage M, Gillespie C, Isasi CR, Jimenez MC, Jordan LC, Judd SE, Lackland D, Lichtman JH, Lisabeth L, Liu S, Longenecker CT, Lutsey PL, Mackey JS, Matchar DB, Matsushita K, Mussolino ME, Nasir K, O'Flaherty M, Palaniappan LP, Pandey A, Pandey DK, Reeves MJ, Ritchey MD, Rodriguez CJ, Roth GA, Rosamond WD, Sampson UKA, Satou GM, Shah SH, Spartano NL, Tirschwell DL, Tsao CW, Voeks JH, Willey JZ, Wilkins JT, Wu JH, Alger HM, Wong SS, Muntner P; American Heart Association Council on Epidemiology and Prevention Statistics Committee and Stroke Statistics Subcommittee. Heart Disease and Stroke Statistics-2018 Update: A Report From the American Heart Association. Circulation. 2018 Mar 20;137(12):e67-e492. doi: 10.1161/CIR.0000000000000558. Epub 2018 Jan 31. No abstract available. PMID 29386200
- [Background] Saran R, Robinson B, Abbott KC, Agodoa LYC, Bhave N, Bragg-Gresham J, Balkrishnan R, Dietrich X, Eckard A, Eggers PW, Gaipov A, Gillen D, Gipson D, Hailpern SM, Hall YN, Han Y, He K, Herman W, Heung M, Hirth RA, Hutton D, Jacobsen SJ, Jin Y, Kalantar-Zadeh K, Kapke A, Kovesdy CP, Lavallee D, Leslie J, McCullough K, Modi Z, Molnar MZ, Montez-Rath M, Moradi H, Morgenstern H, Mukhopadhyay P, Nallamothu B, Nguyen DV, Norris KC, O'Hare AM, Obi Y, Park C, Pearson J, Pisoni R, Potukuchi PK, Rao P, Repeck K, Rhee CM, Schrager J, Schaubel DE, Selewski DT, Shaw SF, Shi JM, Shieu M, Sim JJ, Soohoo M, Steffick D, Streja E, Sumida K, Tamura MK, Tilea A, Tong L, Wang D, Wang M, Woodside KJ, Xin X, Yin M, You AS, Zhou H, Shahinian V. US Renal Data System 2017 Annual Data Report: Epidemiology of Kidney Disease in the United States. Am J Kidney Dis. 2018 Mar;71(3 Suppl 1):A7. doi: 10.1053/j.ajkd.2018.01.002. No abstract available. PMID 29477157
- [Background] Heidenreich PA, Trogdon JG, Khavjou OA, Butler J, Dracup K, Ezekowitz MD, Finkelstein EA, Hong Y, Johnston SC, Khera A, Lloyd-Jones DM, Nelson SA, Nichol G, Orenstein D, Wilson PW, Woo YJ; American Heart Association Advocacy Coordinating Committee; Stroke Council; Council on Cardiovascular Radiology and Intervention; Council on Clinical Cardiology; Council on Epidemiology and Prevention; Council on Arteriosclerosis; Thrombosis and Vascular Biology; Council on Cardiopulmonary; Critical Care; Perioperative and Resuscitation; Council on Cardiovascular Nursing; Council on the Kidney in Cardiovascular Disease; Council on Cardiovascular Surgery and Anesthesia, and Interdisciplinary Council on Quality of Care and Outcomes Research. Forecasting the future of cardiovascular disease in the United States: a policy statement from the American Heart Association. Circulation. 2011 Mar 1;123(8):933-44. doi: 10.1161/CIR.0b013e31820a55f5. Epub 2011 Jan 24. PMID 21262990
- [Background] Ahmed A, Campbell RC. Epidemiology of chronic kidney disease in heart failure. Heart Fail Clin. 2008 Oct;4(4):387-99. doi: 10.1016/j.hfc.2008.03.008. PMID 18760751
- [Background] House AA. Management of Heart Failure in Advancing CKD: Core Curriculum 2018. Am J Kidney Dis. 2018 Aug;72(2):284-295. doi: 10.1053/j.ajkd.2017.12.006. Epub 2018 Feb 23. PMID 29478868
- [Background] Ueda T, Kawakami R, Sugawara Y, Okada S, Nishida T, Onoue K, Soeda T, Okayama S, Takeda Y, Watanabe M, Kawata H, Uemura S, Saito Y. Worsening of renal function during 1 year after hospital discharge is a strong and independent predictor of all-cause mortality in acute decompensated heart failure. J Am Heart Assoc. 2014 Nov 4;3(6):e001174. doi: 10.1161/JAHA.114.001174. PMID 25370599
- [Background] Dries DL, Exner DV, Domanski MJ, Greenberg B, Stevenson LW. The prognostic implications of renal insufficiency in asymptomatic and symptomatic patients with left ventricular systolic dysfunction. J Am Coll Cardiol. 2000 Mar 1;35(3):681-9. doi: 10.1016/s0735-1097(99)00608-7. PMID 10716471
- [Background] Hillege HL, Nitsch D, Pfeffer MA, Swedberg K, McMurray JJ, Yusuf S, Granger CB, Michelson EL, Ostergren J, Cornel JH, de Zeeuw D, Pocock S, van Veldhuisen DJ; Candesartan in Heart Failure: Assessment of Reduction in Mortality and Morbidity (CHARM) Investigators. Renal function as a predictor of outcome in a broad spectrum of patients with heart failure. Circulation. 2006 Feb 7;113(5):671-8. doi: 10.1161/CIRCULATIONAHA.105.580506. PMID 16461840
- [Background] Neal B, Perkovic V, Matthews DR. Canagliflozin and Cardiovascular and Renal Events in Type 2 Diabetes. N Engl J Med. 2017 Nov 23;377(21):2099. doi: 10.1056/NEJMc1712572. No abstract available. PMID 29166232
- [Background] Zinman B, Lachin JM, Inzucchi SE. Empagliflozin, Cardiovascular Outcomes, and Mortality in Type 2 Diabetes. N Engl J Med. 2016 Mar 17;374(11):1094. doi: 10.1056/NEJMc1600827. No abstract available. PMID 26981940
- [Background] Herrington WG, Savarese G, Haynes R, Marx N, Mellbin L, Lund LH, Dendale P, Seferovic P, Rosano G, Staplin N, Baigent C, Cosentino F. Cardiac, renal, and metabolic effects of sodium-glucose co-transporter 2 inhibitors: a position paper from the European Society of Cardiology ad-hoc task force on sodium-glucose co-transporter 2 inhibitors. Eur J Heart Fail. 2021 Aug;23(8):1260-1275. doi: 10.1002/ejhf.2286. Epub 2021 Jul 20. PMID 34184823
- [Background] Verma S, Rawat S, Ho KL, Wagg CS, Zhang L, Teoh H, Dyck JE, Uddin GM, Oudit GY, Mayoux E, Lehrke M, Marx N, Lopaschuk GD. Empagliflozin Increases Cardiac Energy Production in Diabetes: Novel Translational Insights Into the Heart Failure Benefits of SGLT2 Inhibitors. JACC Basic Transl Sci. 2018 Aug 26;3(5):575-587. doi: 10.1016/j.jacbts.2018.07.006. eCollection 2018 Oct. PMID 30456329
- [Background] Mudaliar S, Alloju S, Henry RR. Can a Shift in Fuel Energetics Explain the Beneficial Cardiorenal Outcomes in the EMPA-REG OUTCOME Study? A Unifying Hypothesis. Diabetes Care. 2016 Jul;39(7):1115-22. doi: 10.2337/dc16-0542. PMID 27289124
- [Background] Kumar N, Garg A, Bhatt DL, Sabongui S, Gupta N, Chaudhry S, Arena R, Verma S. Empagliflozin improves cardiorespiratory fitness in type 2 diabetes: translational implications. Can J Physiol Pharmacol. 2018 Nov;96(11):1184-1187. doi: 10.1139/cjpp-2018-0359. PMID 30265814
- [Background] Verma S, Garg A, Yan AT, Gupta AK, Al-Omran M, Sabongui A, Teoh H, Mazer CD, Connelly KA. Effect of Empagliflozin on Left Ventricular Mass and Diastolic Function in Individuals With Diabetes: An Important Clue to the EMPA-REG OUTCOME Trial? Diabetes Care. 2016 Dec;39(12):e212-e213. doi: 10.2337/dc16-1312. Epub 2016 Sep 27. No abstract available. PMID 27679584
- [Background] Bagby SP. Obesity-initiated metabolic syndrome and the kidney: a recipe for chronic kidney disease? J Am Soc Nephrol. 2004 Nov;15(11):2775-91. doi: 10.1097/01.ASN.0000141965.28037.EE. No abstract available. PMID 15504931
- [Background] Smogorzewski M, Piskorska G, Borum PR, Massry SG. Chronic renal failure, parathyroid hormone and fatty acids oxidation in skeletal muscle. Kidney Int. 1988 Feb;33(2):555-60. doi: 10.1038/ki.1988.33. PMID 3361755
- [Background] Rhee EP. Metabolomics and renal disease. Curr Opin Nephrol Hypertens. 2015 Jul;24(4):371-9. doi: 10.1097/MNH.0000000000000136. PMID 26050125
- [Background] Hocher B, Adamski J. Metabolomics for clinical use and research in chronic kidney disease. Nat Rev Nephrol. 2017 May;13(5):269-284. doi: 10.1038/nrneph.2017.30. Epub 2017 Mar 6. PMID 28262773
- [Background] Grams ME, Shafi T, Rhee EP. Metabolomics Research in Chronic Kidney Disease. J Am Soc Nephrol. 2018 Jun;29(6):1588-1590. doi: 10.1681/ASN.2018030256. Epub 2018 May 3. No abstract available. PMID 29724883
- [Background] Kalim S, Rhee EP. An overview of renal metabolomics. Kidney Int. 2017 Jan;91(1):61-69. doi: 10.1016/j.kint.2016.08.021. Epub 2016 Sep 28. PMID 27692817
- [Background] Chen DQ, Cao G, Chen H, Argyopoulos CP, Yu H, Su W, Chen L, Samuels DC, Zhuang S, Bayliss GP, Zhao S, Yu XY, Vaziri ND, Wang M, Liu D, Mao JR, Ma SX, Zhao J, Zhang Y, Shang YQ, Kang H, Ye F, Cheng XH, Li XR, Zhang L, Meng MX, Guo Y, Zhao YY. Identification of serum metabolites associating with chronic kidney disease progression and anti-fibrotic effect of 5-methoxytryptophan. Nat Commun. 2019 Apr 1;10(1):1476. doi: 10.1038/s41467-019-09329-0. PMID 30931940
- [Background] Wang F, Sun L, Sun Q, Liang L, Gao X, Li R, Pan A, Li H, Deng Y, Hu FB, Wu J, Zeng R, Lin X. Associations of Plasma Amino Acid and Acylcarnitine Profiles with Incident Reduced Glomerular Filtration Rate. Clin J Am Soc Nephrol. 2018 Apr 6;13(4):560-568. doi: 10.2215/CJN.07650717. Epub 2018 Mar 8. PMID 29519950
- [Background] Hiltunen TP, Rimpela JM, Mohney RP, Stirdivant SM, Kontula KK. Effects of four different antihypertensive drugs on plasma metabolomic profiles in patients with essential hypertension. PLoS One. 2017 Nov 9;12(11):e0187729. doi: 10.1371/journal.pone.0187729. eCollection 2017. PMID 29121091
- [Background] Cozzolino M, Mangano M, Stucchi A, Ciceri P, Conte F, Galassi A. Cardiovascular disease in dialysis patients. Nephrol Dial Transplant. 2018 Oct 1;33(suppl_3):iii28-iii34. doi: 10.1093/ndt/gfy174. PMID 30281132
- [Background] Zewinger S, Kleber ME, Rohrer L, Lehmann M, Triem S, Jennings RT, Petrakis I, Dressel A, Lepper PM, Scharnagl H, Ritsch A, Thorand B, Heier M, Meisinger C, de Las Heras Gala T, Koenig W, Wagenpfeil S, Schwedhelm E, Boger RH, Laufs U, von Eckardstein A, Landmesser U, Luscher TF, Fliser D, Marz W, Meinitzer A, Speer T. Symmetric dimethylarginine, high-density lipoproteins and cardiovascular disease. Eur Heart J. 2017 May 21;38(20):1597-1607. doi: 10.1093/eurheartj/ehx118. PMID 28379378
- [Background] Potocnjak I, Radulovic B, Degoricija V, Trbusic M, Pregartner G, Berghold A, Meinitzer A, Frank S. Serum concentrations of asymmetric and symmetric dimethylarginine are associated with mortality in acute heart failure patients. Int J Cardiol. 2018 Jun 15;261:109-113. doi: 10.1016/j.ijcard.2018.03.037. Epub 2018 Mar 11. PMID 29550017
- [Background] Schepers E, Barreto DV, Liabeuf S, Glorieux G, Eloot S, Barreto FC, Massy Z, Vanholder R; European Uremic Toxin Work Group (EUTox). Symmetric dimethylarginine as a proinflammatory agent in chronic kidney disease. Clin J Am Soc Nephrol. 2011 Oct;6(10):2374-83. doi: 10.2215/CJN.01720211. Epub 2011 Aug 4. PMID 21817129
- [Background] Memon L, Spasojevic-Kalimanovska V, Stanojevic NB, Kotur-Stevuljevic J, Simic-Ogrizovic S, Giga V, Dopsaj V, Jelic-Ivanovic Z, Spasic S. Are levels of NT-proBNP and SDMA useful to determine diastolic dysfunction in chronic kidney disease and renal transplant patients? J Clin Lab Anal. 2013 Nov;27(6):461-70. doi: 10.1002/jcla.21628. PMID 24218128
- [Background] Daniele G, Xiong J, Solis-Herrera C, Merovci A, Eldor R, Tripathy D, DeFronzo RA, Norton L, Abdul-Ghani M. Dapagliflozin Enhances Fat Oxidation and Ketone Production in Patients With Type 2 Diabetes. Diabetes Care. 2016 Nov;39(11):2036-2041. doi: 10.2337/dc15-2688. Epub 2016 Aug 25. PMID 27561923
- [Background] Ferrannini E, Baldi S, Frascerra S, Astiarraga B, Heise T, Bizzotto R, Mari A, Pieber TR, Muscelli E. Shift to Fatty Substrate Utilization in Response to Sodium-Glucose Cotransporter 2 Inhibition in Subjects Without Diabetes and Patients With Type 2 Diabetes. Diabetes. 2016 May;65(5):1190-5. doi: 10.2337/db15-1356. Epub 2016 Feb 9. PMID 26861783
- [Background] Mulder S, Hammarstedt A, Nagaraj SB, Nair V, Ju W, Hedberg J, Greasley PJ, Eriksson JW, Oscarsson J, Heerspink HJL. A metabolomics-based molecular pathway analysis of how the sodium-glucose co-transporter-2 inhibitor dapagliflozin may slow kidney function decline in patients with diabetes. Diabetes Obes Metab. 2020 Jul;22(7):1157-1166. doi: 10.1111/dom.14018. Epub 2020 Mar 25. PMID 32115853
- [Background] Kappel BA, Lehrke M, Schutt K, Artati A, Adamski J, Lebherz C, Marx N. Effect of Empagliflozin on the Metabolic Signature of Patients With Type 2 Diabetes Mellitus and Cardiovascular Disease. Circulation. 2017 Sep 5;136(10):969-972. doi: 10.1161/CIRCULATIONAHA.117.029166. No abstract available. PMID 28874423
- [Background] Radholm K, Figtree G, Perkovic V, Solomon SD, Mahaffey KW, de Zeeuw D, Fulcher G, Barrett TD, Shaw W, Desai M, Matthews DR, Neal B. Canagliflozin and Heart Failure in Type 2 Diabetes Mellitus: Results From the CANVAS Program. Circulation. 2018 Jul 31;138(5):458-468. doi: 10.1161/CIRCULATIONAHA.118.034222. PMID 29526832
- [Background] Mahaffey KW, Neal B, Perkovic V, de Zeeuw D, Fulcher G, Erondu N, Shaw W, Fabbrini E, Sun T, Li Q, Desai M, Matthews DR; CANVAS Program Collaborative Group. Canagliflozin for Primary and Secondary Prevention of Cardiovascular Events: Results From the CANVAS Program (Canagliflozin Cardiovascular Assessment Study). Circulation. 2018 Jan 23;137(4):323-334. doi: 10.1161/CIRCULATIONAHA.117.032038. Epub 2017 Nov 13. PMID 29133604
- [Background] Zamani P, Rawat D, Shiva-Kumar P, Geraci S, Bhuva R, Konda P, Doulias PT, Ischiropoulos H, Townsend RR, Margulies KB, Cappola TP, Poole DC, Chirinos JA. Effect of inorganic nitrate on exercise capacity in heart failure with preserved ejection fraction. Circulation. 2015 Jan 27;131(4):371-80; discussion 380. doi: 10.1161/CIRCULATIONAHA.114.012957. Epub 2014 Dec 22. PMID 25533966
- [Background] Chong J, Soufan O, Li C, Caraus I, Li S, Bourque G, Wishart DS, Xia J. MetaboAnalyst 4.0: towards more transparent and integrative metabolomics analysis. Nucleic Acids Res. 2018 Jul 2;46(W1):W486-W494. doi: 10.1093/nar/gky310. PMID 29762782
- See also: Reference #28 in protocol. Symmetric and asymmetric dimethylarginine as risk markers of cardiovascular disease, all-cause mortality and deterioration in kidney function in persons with type 2 diabetes and microalbuminuria. — https://cardiab.biomedcentral.com/articles/10.1186/s12933-017-0569-8